CLINICAL TRIAL: NCT00003829
Title: A Phase II Study of Alternating Cycles of Fludarabine and Cyclophosphamide in Previously Untreated Patients With B-cell CLL
Brief Title: Chemotherapy in Treating Patients With Previously Untreated Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-978151; NCCTG-978151; CDR0000066985 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02296 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fludarabine + cyclophosphamide (Experimental): Patients receive alternating courses of fludarabine and cyclophosphamide. Fludarabine is administered IV over 10-30 minutes on days 1-5 of courses 1, 3, and 5. Cyclophosphamide is administered IV over 30-60 minutes on day 1 of courses 2, 4, and 6. Treatment repeats every 4 weeks. Patients achieving clinical complete remission (CCR) after 6 courses of chemotherapy receive 2 additional courses (one course of each drug). Patients achieving partial remission after 6 courses of chemotherapy also receive 2 additional courses. If these patients then achieve CCR, they receive another 2 courses. Patients are followed every 3 months.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Alternating treatment with more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of fludarabine alternating with cyclophosphamide in treating patients who have previously untreated chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rate and duration of complete and partial remissions in patients with previously untreated B-cell chronic lymphocytic leukemia after treatment with alternating courses of fludarabine and cyclophosphamide. II. Monitor and assess toxicity of this regimen in these patients. III. Utilize molecular genetic studies and flow cytometry on peripheral blood cells from patients achieving complete remission by conventional criteria. IV. Apply FISH techniques using probes to chromosomes 12 and 13 as prognostic factors for time to progression and overall survival of these patients.

OUTLINE: Patients receive alternating courses of fludarabine and cyclophosphamide. Fludarabine is administered IV over 10-30 minutes on days 1-5 of courses 1, 3, and 5. Cyclophosphamide is administered IV over 30-60 minutes on day 1 of courses 2, 4, and 6. Treatment repeats every 4 weeks. Patients achieving clinical complete remission (CCR) after 6 courses of chemotherapy receive 2 additional courses (one course of each drug). Patients achieving partial remission after 6 courses of chemotherapy also receive 2 additional courses. If these patients then achieve CCR, they receive another 2 courses. Patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of B-cell chronic lymphocytic leukemia (CLL) manifested by all of the following: Threshold peripheral lymphocyte count greater than 5000/mm3 Small to moderate peripheral lymphocytes with no greater than 55% prolymphocytes Peripheral lymphocyte count less than 15,000/mm3 At least 30% lymphoid cells in bone marrow Monoclonality of B lymphocytes Active disease by at least one of the following criteria: Weight loss of at least 10% within the past 6 months or prolonged fever or night sweats without evidence of infection Progressive marrow failure (stage III or IV disease) manifested by Hemoglobin less than 11 g/dL (anemia) AND/OR Platelet count less than 100,000/mm3 (thrombocytopenia) Autoimmune anemia and/or thrombocytopenia minimally responsive to corticosteroid therapy Massive or progressive splenomegaly Massive or progressive lymphadenopathy Progressive lymphocytosis (not due to the effects of corticosteroids) Marked hypogammaglobulinemia or development of monoclonal protein in the absence of any of the above criteria is not sufficient for eligibility

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 1.5 times ULN (unless due to hemolysis or CLL) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No New York Heart Association class III or IV heart disease No myocardial infarction in the past month Other: No uncontrolled infection No active infection with HIV (AIDS) No other malignancy within past 2 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior interferon allowed Chemotherapy: No prior cytotoxic chemotherapy Endocrine therapy: See Disease Characteristics Prior corticosteroids, somatostatin analogues, and tamoxifen allowed Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 1999-08; Primary Completion 2001-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
proportion of confirmed responses | Up to 6 months

SECONDARY OUTCOMES:
overall survival | Up to 5 years
progression free survival | Up to 5 years
time to progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic
Locations (17):
- United States (17):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota